CLINICAL TRIAL: NCT03110952
Title: A Phase 1, Randomized, Placebo-Controlled, Observer-Blind, Single-Center, Study of TDENV-PIV and TDENV-F17 Dengue Vaccine Platforms in a Heterologous Prime Boost Strategy in Healthy Adults in a Non-Endemic Region
Brief Title: TDENV PIV and LAV Dengue Prime-boost Strategy Using AS03B Adjuvant
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of materials, not moving forward
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S-14-08; DPIV-020 (Other: Sponsor); 201126 (Other: GSK eTrack)
Record Dates: First submitted 2015-04-28; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue | interventions — Serogroup; Vaccines, Attenuated; Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- TDENV-PIV x2 (Experimental): 2 doses of TDENV-PIV on Day 0 and Day 28
  Interventions: Biological: TDENV-PIV
- TDENV-F17/TDENV-PIV (Experimental): 1 dose TDENV-F17 on Day 0 and 1 dose TDENV-PIV on Day 28
  Interventions: Biological: TDENV-PIV; Biological: TDENV-F17
- TDENV-PIV/TDENV-F17 (Experimental): 1 dose TDENV-PIV on Day 0 and 1 dose TDENV-F17 on Day 28
  Interventions: Biological: TDENV-PIV; Biological: TDENV-F17
- Placebo (Placebo Comparator): 2 doses placebo (phosphate buffered saline) Day 0 and Day 28
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: TDENV-PIV — Single-dose vial with pre-filled syringe, subcutaneous injection
  Other Names: Tetravalent dengue virus, purified inactivated vaccine, TDENV-PIV with AS03B adjuvant; Inactivated dengue virus types 1-4 (1 µg/serotype) with AS03B adjuvant
  Arms: TDENV-F17/TDENV-PIV; TDENV-PIV x2; TDENV-PIV/TDENV-F17
Biological: TDENV-F17 — Single-dose vial with pre-filled syringe 0.5 mL administered intramuscularly
  Other Names: Tetravalent dengue virus, live, attenuated vaccine, TDENV-F17; Live attenuated dengue virus types 1-4
  Arms: TDENV-F17/TDENV-PIV; TDENV-PIV/TDENV-F17
Other: Placebo — 0.5 mL vial
  Other Names: Placebo, sterile phosphate-buffered saline solution for injection
  Arms: Placebo

SUMMARY:
The potential synergistic effect of administering 2 dengue vaccine candidates that were previously shown to be safe and immunogenic in humans will be evaluated in this study. A prime-boost study of tetravalent dengue virus purified inactivated vaccine (TDENV-PIV) with the GSK AS03B adjuvant and tetravalent dengue live attenuated virus (TDENV-LAV) vaccine Formulation 17 (F17) will gather data to help better understand the human immune response to dengue vaccination and infection.

This study is being done to evaluate the safety and immune reaction of administering one dose of dengue purified inactivated vaccine and one dose of dengue live attenuated vaccine compared to two doses of inactivated vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., document events in memory aid, return for follow-up visits, etc.)
* Between 18 and 39 years of age (inclusive) at the time of consent
* Written informed consent obtained from the subject
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines/placebo during the period starting 30 days preceding the first dose of study vaccine/placebo and/or planned use during the study period
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 180 days prior to the first vaccine/placebo dose (for corticosteroids, this will mean prednisone 20 mg/day or equivalent; inhaled and topical steroids are allowed)
* Planned administration or administration of a vaccine/product not foreseen by the study protocol during the period starting 30 days before or after each scheduled dose of an investigational product or placebo.
* Planned administration of any flavivirus vaccine for the entire study duration
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or an approved/cleared non-investigational product (pharmaceutical product or device).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency
* History and family history of a bleeding disorder
* History of past flavivirus infection or vaccination (Yellow Fever, tick-borne encephalitis virus (TBEV), Japanese encephalitis virus (JEV), West Nile virus (WNV), dengue (DENV)
* History of, or current, auto-immune disease
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine/placebo or related to a study procedure
* Major congenital defects or serious chronic illness
* History of any neurological disorders or seizures
* Acute disease and/or fever (≥ 100.4° ◦F / 38.0° ◦C, oral body temperature) at the time of enrollment (a subject with a minor illness, i.e., mild diarrhea, mild upper respiratory infection, etc., without fever, may be enrolled at the discretion of the investigator)
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by physical examination or laboratory screening tests
* Administration of immunoglobulins and/or any blood products during the period starting 90 days preceding the first dose of study vaccine/placebo or planned administration during the study period
* History of chronic alcohol consumption and/or drug abuse
* A planned move to a location that will prohibit participating in the trial until study end for the participant
* Any other condition which, in the opinion of the investigator, prevents the subject from participating in the study.
* Subject seropositive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), or human immunodeficiency virus antibodies (anti-HIV)
* Safety laboratory test results that are outside the acceptable values at screening.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Number of and intensity of solicited local and general adverse events (AEs) during the 7-day follow-up period after each vaccination | Day 7 and Day 35
Number of and intensity of unsolicited adverse events (AEs) during the 7-day follow-up period after each vaccination | Day 7 and Day 35
Number of serious adverse events (SAEs) | Day 35
Number of potential immune-mediated diseases (pIMDs) and medicall attended AEs | Day 56
Geometric mean titers (GMTs) of neutralizing antibodies to each DENV serotype | Day 56
  Assessment of neutralizing antibodies against DENV type 1-4 will be performed by a validated microneutralizing antibody assay.
Number of participants seropositive for each DENV serotype | Day 56
  Seropositive will be determined by 50% reduction in viral infection (MN50)
Number of participants trivalent and tetravalent seropositive | Day 56
  Seropositive will be determined by 50% reduction in viral infection (MN50)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Polhemus, Principal Investigator — Upstate Medical University, SUNY
Locations (1):
- Upstate Medical University, SUNY, Syracuse, New York, United States